CLINICAL TRIAL: NCT00083720
Title: A Phase II Multicenter Study of Erbitux (Cetuximab) in Patients With Refractory, EGFR-Negative Metastatic Colorectal Carcinoma
Brief Title: Erbitux (Cetuximab) Given Alone to Patients With EGFR-Negative Metastatic Colon or Rectal Cancer That is Refractory to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP02-0451
Record Dates: First submitted 2004-05-28; First posted 2004-06-02 (Estimated); Results first posted 2009-10-23 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Colorectal Neoplasms; Metastases; Neoplasm
Keywords: EGFR-undetectable; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cetuximab (Experimental): Initial dose of 400 mg/m2 intravenously (i.v.) over 120 minutes, followed by 250 mg/m2 weekly i.v. over 60 minutes
  Interventions: Biological: cetuximab

INTERVENTIONS:
Biological: cetuximab — Initial dose of 400 mg/m2 intravenously (i.v.) over 120 minutes, followed by 250 mg/m2 weekly i.v. over 60 minutes
  Other Names: Erbitux™

SUMMARY:
This is a phase II, multicenter, open-label study of cetuximab in patients with epidermal growth factor receptor (EGFR) negative, metastatic colorectal carcinoma who have progressed after receiving at least one standard chemotherapeutic regimen that included a fluoropyrimidine. Target enrollment is 80 evaluable patients.

Patients with EGFR-negative metastatic colorectal carcinoma who have progressed after receiving at least one standard chemotherapeutic regimen that included a fluoropyrimidine, will receive an initial dose of cetuximab, 400 mg/m2 , intravenously (i.v.) over 120 minutes, followed by weekly treatment with cetuximab, 250 mg/m2 i.v. over 60 minutes. Patients who experience unacceptable toxicity or who have progressive disease (PD) will not receive further cetuximab therapy.

Patients will be evaluated for a tumor response at a minimum of every 6 weeks while on cetuximab therapy. Patients with stable disease (SD), partial response (PR), or a complete response (CR) may continue to receive weekly cetuximab therapy, unless they are dose-delayed or discontinued because of toxicity. Patients who have a PR or CR must have a confirmatory tumor assessment no less than 4 weeks after the initial evaluation demonstrating a response. To evaluate the objective response rate, a single-stage design will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed written informed consent.
* Histologically- or pathologically- confirmed metastatic colorectal carcinoma;
* Documented PD after treatment with at least one standard chemotherapy regimen for metastatic colorectal carcinoma;
* The chemotherapy regimen on which the patient progressed, must have included a fluoropyrimidine;
* Bidimensionally measurable disease;
* Immunohistochemical evidence of an absence of EGFR expression, (ie, EGFR-negative). Patients who do not have tumor tissue available for EGFR testing will undergo biopsy of accessible tumor. A reference laboratory designated by ImClone will perform the EGFR assay.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1 at study entry;
* Adequate recovery from recent surgery, chemotherapy, and radiation therapy. At least 30 days must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or medical device, or prior radiation therapy;
* Accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center.
* Men and women, 18 years of age and older

Exclusion Criteria:

* Women of child bearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to cetuximab administration.
* Sexually active fertile men not using effective birth control.
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent;
* A serious uncontrolled medical disorder that would impair the ability of the patient to receive protocol therapy;
* A history of uncontrolled angina, arrhythmias or congestive heart failure;
* Symptomatic or uncontrolled metastases to the central nervous system. Patients receiving a glucocorticoid for central nervous system (CNS) metastases will be excluded, but those receiving anticonvulsants will be eligible.
* Any concurrent malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix. Patients with a previous malignancy but without evidence of disease for greater than or equal to 5 years will be allowed to enter the trial;
* Inadequate hematologic function defined by an absolute neutrophil count (ANC) less than 1,500/mm3 , a platelet count less than 100,000/mm3 , or a hemoglobin level less than 9 g/dL.
* Inadequate hepatic function, defined by a total bilirubin level greater than or equal to 1.5 times the upper limit of normal (ULN) and aspartate transaminase (AST) or alanine transaminase (ALT) levels greater than or equal to 5.0 times the ULN.
* Inadequate renal function defined by a serum creatinine level greater than 1.5 times the ULN.
* Prior cetuximab or other therapy, which specifically and directly targets the EGF pathway.
* Prior hypersensitivity reaction to chimerized or murine monoclonal antibody therapy.
* Any chemotherapy not indicated in the study protocol, radiation therapy, hormonal therapy (except for physiological replacement), or any other investigational agent.
* Prisoners or patients who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious disease) illness.
* Employees of the investigator or study center with direct involvement in this study or other studies under the direction of the investigator or study center, as well as family members of the employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (26):
- United States (23):
  - ImClone Investigational Site, Campbell, California
  - ImClone Investigational Site, Los Angeles, California
  - ImClone Investigational Site, Soquel, California
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Ormond Beach, Florida
  - ImClone Investigational Site, Gurnee, Illinois
  - ImClone Investigational Site, Evansville, Indiana
  - ImClone Investigational Site, Indianapolis, Indiana
  - ImClone Investigational Site, Lexington, Kentucky
  - ImClone Investigational Site, Louisville, Kentucky
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Ann Arbor, Michigan
  - ImClone Investigational Site, Kalamazoo, Michigan
  - ImClone Investigational Site, St Louis, Missouri
  - ImClone Investigational Site, Armonk, New York
  - ImClone Investigational Site, East Setauket, New York
  - ImClone Investigational Site, Durham, North Carolina
  - ImClone Investigational Site, Sellingsgrove, Pennsylvania
  - ImClone Investigational Site, Arlington, Texas
  - ImClone Investigational Site, Bryan, Texas
  - ImClone Investigational Site, Temple, Texas
- Canada (3):
  - ImClone Investigational Site, Oshawa, Ontario
  - ImClone Investigational Site, Ottawa, Ontario
  - ImClone Investigational Site, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 87 patients were enrolled between 22 Oct 2004 and 20 Aug 2007 at nine sites in the USA and four sites in Canada.
Groups:
- Cetuximab: Initial dose of 400 mg/m2 i.v. over 120 minutes, followed by 250 mg/m2 weekly i.v. over 60 minutes
Period: Overall Study
Arm/Group | Cetuximab
Started | 85 (Patients analyzed for efficacy who met the epidermal growth factor receptor (EGFR) negative criteria)
Completed | 85 (Two patients died prior to receiving cetuximab.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 59
Region of Enrollment [Number; unit: participants]
  United States | 20
  Canada | 65

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Overall Resonse
Description: Determine the response rate (complete response [CR] and partial response [PR]) in patients with epidermal growth factor receptor (EGFR)-negative metastatic colorectal carcinoma treated with cetuximab, as classified by the investigator according to the World Health Organization (WHO) criteria. The calculation was the total number of patients with CR or PR divided by the total number of patients treated.
Time Frame: Tumor evaluations were performed at a minimum every 6 weeks while on cetuximab therapy until progressive disease (PD) or recurrence. Patients with a PR or CR had a confirmatory tumor assessment no less than 4 weeks after the initial evaluation.
Population: The overall response rate was calculated for the modified Intent to Treat (mITT) population.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 85
percentage of participants | 8.2 [3.4 to 16.2]

2. Secondary Outcome: Percentage of Participants With Disease Control (CR, PR, or SD)
Description: This is the total number of patients with a best overall response of CR, PR, and stable disease (SD) divided by the total number of patients treated.
Time Frame: Tumor evaluations were performed at a minimum of every 6 weeks while on cetuximab therapy. Patients with a PR or CR had a confirmatory tumor assessment no less than 4 weeks after the initial evaluation demonstrating a response.
Population: Disease control rate was the total number of patients with best overall response of CR, PR and SD divided by the total number of patients treated.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 85
Percentage of participants | 49.4 [38.4 to 60.5]

3. Secondary Outcome: Duration of Response
Description: In patients with a best overall response of CR or PR, the duration of response is measured from the date criteria are first met for CR or PR, until the first date that Progressive Disease (PD) is objectively documented or death occurs. Duration of response of living patients with no evidence of PD was censored on the date of their last tumor assessment.
Time Frame: The duration of response was measured from the date of response to the first date of PD (range 2 to 7 months).
Population: The duration of response was calculated for the subgroup of the mITT population who demonstrated a response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab
Number analyzed (Participants) | 7
Months | 5.1 [2.7 to 6.9]

4. Secondary Outcome: Time to Progression
Description: This measure was defined as the time from the first day of treatment until the date of PD. Deaths without objective progression were censored. Patients who did not progress were censored at their last day of tumor assessment.
Time Frame: Patients with PD after receiving at least one standard chemotherapeutic regimen that included a fluoropyrimidine (range: 1-3 months).
Population: This measure was calculated for the mITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab
Number analyzed (Participants) | 85
Months | 2.5 [1.3 to 2.8]

5. Secondary Outcome: Overall Survival
Description: This measure is defined as the time from the first day of therapy to the date of death. Survival of living patients or those lost to follow-up were censored on the last date the patients were known to be alive.
Time Frame: Survival information was collected every 3 months after completion of therapy and/or follow-up up to 24 months.
Population: Overall survival was calculated from the time of the first day of therapy to the date of death for the mITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab
Number analyzed (Participants) | 85
Months | 10.0 [7.5 to 12.0]

6. Primary Outcome: Number of Participants With Adverse Events
Description: Reported adverse events (AEs) per patient were coded according to the corresponding preferred term and system organ class in the Medical Dictionary for Regulatory Activities dictionary. The National Cancer Insititute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3.0 was used to grade all AEs. The collection of AEs began at the time the patient received the first cetuximab dose and continued during the study until 30 days after the last dose of cetuximab. All patients who were enrolled and treated with cetuximab were assessed for safety (mITT population, as treated).
Time Frame: An adverse event (AE) was included in the safety analysis if its onset date occurred anytime during cetuximab treatment or up to 30 days after the last dose of cetuximab.
Population: Patients who were enrolled and treated with any quantity of cetuximab constitute the mITT population. Since this trial was a single arm trial, the mITT population used for the efficacy analyses was also used for the safety analyses.
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 85
Participants | 85

7. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Reported SAEs per patient were coded according to the corresponding preferred term and system organ class in the Medical Dictionary for Regulatory Activities. The NCI-CTCAE Version 3.0 was used to grade all SAEs. An SAE was any untoward medical occurrence that resulted in death, persistent/significant disability/incapacity, was life threatening, required inpatient hospitalization or caused prolongation of existing hospitalization,congenital anomaly/birth defect, or any important medical event.
Time Frame: A serious adverse event (SAE) was included in the safety analysis if its onset date occurred anytime during cetuximab treatment or up to 30 days after the last dose of cetuximab.
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 85
Participants | 19

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time that the patient received the initial cetuximab infusion and continued during the study until 30 days after the last dose of cetuximab.
Description: The NCI-CTCAE V3.0 toxicity criteria was used to grading the severity of all AEs.
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 19/85
Other Adverse Events (participants affected / at risk) | 84/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (N=85)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 3 (3)
Death (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dissociation (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab (N=85)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 8 (11)
Diarrhea (Gastrointestinal disorders) | 12 (17)
Nausea (Gastrointestinal disorders) | 13 (14)
Stomatitis (Gastrointestinal disorders) | 9 (10)
Vomiting (Gastrointestinal disorders) | 8 (11)
Chills (General disorders) | 6 (8)
Fatigue (General disorders) | 27 (33)
Oedema peripheral (General disorders) | 6 (6)
Pyrexia (General disorders) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 20 (21)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Headache (Nervous system disorders) | 25 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 73 (102)
Dry skin (Skin and subcutaneous tissue disorders) | 15 (16)
Nail disorder (Skin and subcutaneous tissue disorders) | 9 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
Skin disorder (Skin and subcutaneous tissue disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may not independently publish/disclose any study data, findings or conclusions except as part of an overall multi-center publication. After final publication, or if a draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to review for sponsor confidential information which may be redacted at sponsor request. Publication may be delayed up to 90 days to seek patent protection.